CLINICAL TRIAL: NCT03429634
Title: Comparative Study of Balloon-Stent Kissing Technique Versus Jailed Wire Technique for the Interventional Treatment of Coronary Bifurcation Lesions
Brief Title: Balloon-Stent Kissing Technique Versus Jailed Wire Technique for the Coronary Bifurcation Lesions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dalian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DalianU
Record Dates: First submitted 2018-01-04; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Balloon-Stent Kissing technique (Experimental): randomly, patients with bifurcation lesion treated by Balloon-Stent Kissing intervention technique in this group.For procedure,stent in main vessel and balloon protect of side branch,final kiss-balloon was performed.
  Interventions: Procedure: Balloon-Stent Kissing technique; Procedure: Jailed Wire technique
- Jailed Wire technique (Sham Comparator): randomly,patients with bifurcation lesion treated by Jailed Wire intervention technique in this group.For procedure,stent in main vessel and only wire protect of side branch.If need,post-stent rewire of branch,and balloon dilation of side branch was performed.
  Interventions: Procedure: Balloon-Stent Kissing technique; Procedure: Jailed Wire technique

INTERVENTIONS:
Procedure: Balloon-Stent Kissing technique — All patients underwent coronary angiogram that confirmed true bifurcation lesions, and received PCI treatment,Balloon-Stent Kissing Technique (BSKT)for the interventional treatment of coronary bifurcation lesion
Procedure: Jailed Wire technique — All patients underwent coronary angiogram that confirmed true bifurcation lesions, and received PCI treatment, Jailed Wire technique(JWT) for the interventional treatment of coronary bifurcation lesion

SUMMARY:
To compare the immediate and long-term clinical outcomes between Balloon-Stent Kissing Technique (BSKT) and Jailed Wire Technique (JWT) for the interventional treatment of coronary bifurcation lesions.

DETAILED DESCRIPTION:
Coronary bifurcation lesions account for 15-20% of percutaneous coronary interventions (PCIs)[1-2]. They have lower success rate after operation, higher re-stricture ratio by radiography and frequent complications, which result in adverse clinical outcomes as compared to non-bifurcation lesions[3-5]. Secure and efficient treatment strategies for PCI and bifurcation lesions are research hotspots for cardiovascular surgeons. Single-side stand strategy (main-support implantation stand or side-support implantation stand when necessary) is currently preferred for bifurcation lesions[2,6]. However, as main-support implantation stand could lead to plaque transposition, bifurcation ridge excursion and side a sandwich, the side openings could become narrower or even blocked[7]. In 2011, our centre initiated the use of balloon-stent kissing technique (BSKT)[8] to protect the side branch, which has higher success rate after operation, lower block ratio of side branch and lower incidence of perioperative adverse events, which led to immediate clinical effect. This study compared BSKT versus Jailed Wire Technique (JWT) in the interventional treatment of coronary bifurcation lesions to further clarify BSKT's efficacy and advantages.

ELIGIBILITY:
Inclusion Criteria:

* 1. patients with CHD; 2. coronary arteriography revealed true bifurcation lesion

Exclusion Criteria:

* 1. severe carcified lesion; 2. left main lesion; 3. severe heart failure(NYHA grade 4)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Perioperative major adverse cardiovascular (MACE) events （%） | up to 72hr after PCI
  total percent of cardiac death, perioperative myocardial infarction and target lesion revascularization

SECONDARY OUTCOMES:
long-term clinical outcomes（%） | post-PCI to mean 19 month follow up
  total percent of angina pectoris, CCS classification ≥Ⅱ level and severe heart failure (NYHA class),cardiac death, perioperative myocardial infarction and target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: zhenguo Zheng, Dr., Study Director — zhongshan Hospital affiliated to dalian University
Locations (1):
- Dept. of Cardiology, Affiliated Zhongshan hospital of Dalian University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lassen JF, Holm NR, Stankovic G, Lefevre T, Chieffo A, Hildick-Smith D, Pan M, Darremont O, Albiero R, Ferenc M, Louvard Y. Percutaneous coronary intervention for coronary bifurcation disease: consensus from the first 10 years of the European Bifurcation Club meetings. EuroIntervention. 2014 Sep;10(5):545-60. doi: 10.4244/EIJV10I5A97. PMID 25256198
- See also: Consensus Development Conference — http://www.ncbi.nlm.nih.gov